CLINICAL TRIAL: NCT05308043
Title: Deep Learning Computer-aided Detection System for Retinoblastoma Detection and Monitoring.
Brief Title: Deep Learning in Retinoblastoma Detection and Monitoring.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Wenbin Wei, Prof., Beijing Tongren Hospital
Other Study IDs: AI in retinoblastoma
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinoblastoma patients: Retinoblastoma patients who undergo standard medical care in Beijing Tongren Hospital. The anonymous image of these patients will be prospectively collected and labelled by senior ophthalmologists.
  Interventions: Diagnostic Test: Deep learning algorism

INTERVENTIONS:
Diagnostic Test: Deep learning algorism — A deep learning algorism that was developed previous would be applied to identify retinoblastoma tumours on Retcam images and distinguish between active and inactive retinoblastoma tumours. The decision of two different senior ophthalmologists would be the gold standard.

SUMMARY:
Retinoblastoma is the most common eye cancer of childhood. Eye-preserving therapies require routine monitoring of retinoblastoma regression and recurrence to guide corresponding treatment. In the current study, we develop a deep learning algorism that can simultaneously identify retinoblastoma tumours on Retcam images and distinguish between active and inactive retinoblastoma tumours. This algorism will be validated through a prospectively collected dataset.

DETAILED DESCRIPTION:
Retinoblastoma, the most common eye cancer of childhood, affects 1 in 15 000 to 1 in 18 000 live births. China has the second-largest number of patients with retinoblastoma in the world. Eye-preserving therapies have been used widely in China for approximately 15 years. Eye-preserving therapies require routine monitoring of retinoblastoma regression and recurrence to guide corresponding treatment. However, the major amount of qualified ophthalmologists are concentrated in several medical centres. Deep learning based on Retcam examination that can identify retinoblastoma will reduce screening accuracy of the local hospitals and reduce monitoring wordload. In the current study, a deep learning algorism was developed that can simultaneously identify retinoblastoma tumours on Retcam images and distinguish between active and inactive retinoblastoma tumours. This algorism will be validated through a prospectively collected dataset.

ELIGIBILITY:
Inclusion Criteria:

* Retinoblastoma patients undergo standard medical management.

Exclusion Criteria:

* The operators identified images non-assessable for a correct diagnosis, due to reasons such as blur and defocus, and excluded them from further analysis.

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Retinoblastoma patients undergo standard medical management.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis accurcy of deep learning algorism | 1 week
  The diagnosic accurcy of this deep learning algorism is the proportion of true positive and true negative in all evaluated cases

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Bin Wei, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang R, Dong L, Li R, Zhang K, Li Y, Zhao H, Shi J, Ge X, Xu X, Jiang L, Shi X, Zhang C, Zhou W, Xu L, Wu H, Li H, Yu C, Li J, Ma J, Wei W. Automatic retinoblastoma screening and surveillance using deep learning. Br J Cancer. 2023 Aug;129(3):466-474. doi: 10.1038/s41416-023-02320-z. Epub 2023 Jun 21. PMID 37344582